CLINICAL TRIAL: NCT03806231
Title: A Trial of Cervidil (Dinoprostone, Prostaglandin E2 (PGE2), Insert) for Outpatient Pre-induction of Cervical Ripening in Women at 39.0-41.6 Weeks Gestation
Brief Title: A Trial of Cervidil for Outpatient Pre-induction of Cervical Ripening
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor declined to provide further funding/product support.
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OutpatientCervidilTrial
Record Dates: First submitted 2018-10-25; First posted 2019-01-16 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: Cervical Ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Outpatient Cervical Ripening (Experimental): Patients randomized to the outpatient cervical ripening arm will come in for a scheduled visit in Labor and Delivery prior to her scheduled induction. A research nurse will examine her and place the Cervidil insert into the posterior vaginal fornix. The patient will be monitored for 2 hours and sent home after a the following are present: (1) reactive non-stress test (NST) (2) category 1 tracing x 2 hours (3) no vaginal bleeding (4) normal maternal vital signes (5) intact bag of water (BOW) and (6) less than 1 contraction every 10 minutes at the time of discharge. The patient will remove the insert the following morning prior to her scheduled induction.
  Interventions: Drug: Outpatient Dinoprostone 10mg
- Inpatient Cervical Ripening (Active Comparator): The patient will be admitted into the Labor and Delivery unit prior to her scheduled induction. A research nurse will examine her and place the Cervidil insert into the posterior vaginal fornix. The patient will be watched with continuous fetal monitoring for 2 hours. The patient remains hospitalized and the following morning the induction will be started per Intermountain Healthcare protocol.
  Interventions: Drug: Inpatient Dinoprostone 10 mg

INTERVENTIONS:
Drug: Outpatient Dinoprostone 10mg — Dinoprostone (10 mg) is a vaginal insert approved to start and/or continue the ripening of the cervix in pregnant women who are at or near the time of delivery and in whom there is a medical reason for inducing (bringing on) labor. Women randomized to the outpatient cervical ripening group will be administered the drug prior to their induction and discharged after monitoring and physician approval. They will return for their schedule induction.
  Other Names: Outpatient Cervidil
  Arms: Outpatient Cervical Ripening
Drug: Inpatient Dinoprostone 10 mg — Dinoprostone (10 mg) is a vaginal insert approved to start and/or continue the ripening of the cervix in pregnant women who are at or near the time of delivery and in whom there is a medical reason for inducing (bringing on) labor. Women who are randomized to the inpatient cervical ripening group will be administered the drug prior to their induction and remain hospitalized.
  Other Names: Inpatient Cervidil
  Arms: Inpatient Cervical Ripening

SUMMARY:
Induction of labor is a frequently planned obstetric procedure. Induction for women with an unfavorable cervix (bishop score <6) increases the risk of cesarean section. This risk may be reduced by ripening or softening the cervix before the induction of labor. This protocol outlines a randomized trial of 200 women evaluating the placement and use of Cervidil to the post vaginal fornix to soften the cervix in preparation for induction.

This trial is looking at inpatient vs outpatient pre-induction cervical ripening using Cervidil and the effects on (1) maternal and newborn outcomes including time of admission to delivery, (2) system healthcare cost, (3) cost to patient, and (4) patient satisfaction.

The investigators hypothesize when compared to patients admitted to the hospital for cervical ripening:

1. From the time of admission, patients in the outpatient cervical ripening arm will progress to complete cervical dilation in less time.
2. The total overall cost of care for the encounter will be reduced for the group in the outpatient cervical ripening arm.
3. Patients in the outpatient cervical ripening arm will have more overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Accurate gestational age dating by Intermountain dating criteria placing the patient between 39 0/7 and 41 6/7 weeks gestational at time of cervical ripening
* Planning to undergo cervical ripening for induction of labor
* Participants must live <20 minutes away from the enrolling facility, or must stay < 20 minutes away.
* Pregnant women between the ages of 18 and 41 at the time of enrollment.
* Fetus in vertex position

Exclusion Criteria:

* Gestational age < 39 weeks or > 41 weeks and 6 days
* Hypertension (chronic, transitional, gestational, preeclampsia)
* Multiple gestation
* Intrauterine Growth Restriction
* Anticoagulant therapy or at high risk for thromboembolism
* Cardiac disease other than class I per American Heart Association (AHA)
* Prior incision in the contractile portion of the uterus
* Placenta previa
* Oligohydramnios per American College of Obstetricians and Gynecologists (ACOG) criteria: AFI < 5 or deepest vertical pocket <= 2
* Polyhydramnios per ACOG criteria: Amniotic Fluid Index (AFI) >= 24
* Cervical dilation >= 3cm
* Known fetal anomaly that would require advanced neonatal care
* Pitocin-induction of labor is otherwise contraindicated
* Patient is receiving other uterotonics (e.g. oxytocin, Cytotec, etc.)
* Fetal distress
* Unexplained vaginal bleeding during the pregnancy
* Sensitivity to prostaglandin
* Evidence of or suspicion of marked cephalo-pelvic disproportion (per the Cervidil package insert revision 02/2016, Ferring Pharmaceuticals Inc. Parsippany, NJ)

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nichols, DO, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Dixie Regional Medical Center, St. George, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Started | 4 | 4
Completed | 2 | 4
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 24.5 [18 to 27] | 30.5 [24 to 39] | 27.5 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Dilation Completion Time
Description: Time of admission for induction to complete dilation.
Time Frame: Time of admission to completion of dilation (up to 48 hours)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Total Cost of Induction Charged to Patient
Description: Total hospital charges to patient, as obtained by Intermountain Healthcare billing
Time Frame: Through study completion (up to 1 year)
Population: Trial terminated prior to meeting sample size for sufficient analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Satisfaction: Survey
Description: Measured by patient satisfaction/pain/anxiety survey. Questions about patient satifisfaction, pain, and anxiety will have Likert scale responses that range from 2 to 10 choices. Each question will be evaluated independently between cases and controls.
Time Frame: Time of delivery to discharge (up to 96 hours)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vaginal Delivery Rate
Description: Number of patients enrolled who delivered vaginally
Time Frame: Through study completion (up to 1 year)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Operative Vaginal Delivery Rate
Description: Number of patients enrolled who required an operative vaginal delivery
Time Frame: Through study completion (up to 1 year)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cesarean Delivery Rate
Description: Number of patients enrolled who had a c-section delivery
Time Frame: Through study completion (up to 1 year)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Start of Oxytocin Until Delivery
Description: Length of time between patient receiving oxytocin and delivery
Time Frame: Time oxytocin is administered to time of delivery (up to 24 hours)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time of Delivery Until Discharge
Description: Length of time between delivery and discharge.
Time Frame: Time of delivery to discharge (up to 96 hours)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time of Admission Until Discharge
Description: Total length of time patient was hospitalized, from admission to Labor and Delivery until discharge
Time Frame: Time of admission to labor and delivery to discharge (up to 96 hours)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Infant 5 Minute APGAR Score
Description: APGAR score 5 minutes after delivery. The score ranges from 0 to 10 and a score of 7 or above is considered good health.
Time Frame: From delivery to 5 minutes following delivery
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Time of Admission to Postpartum
Description: Length of stay on postpartum unit.
Time Frame: Time of admission to postpartum until discharge (up to 96 hours)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: NICU Admission
Description: Length of time spent in NICU
Time Frame: Time of admission to NICU to discharge (up to 3 weeks)
Population: Trial terminated prior to meeting sufficient sample size for analysis.
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Enrollment period - Approximately 5 months
Arm/Group | Outpatient Cervical Ripening | Inpatient Cervical Ripening
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Cervical Ripening (N=4) | Inpatient Cervical Ripening (N=4)
Non-Serious Adverse Event (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Post-surgical bleeding

LIMITATIONS AND CAVEATS:
Trial terminated prior to meeting sufficient sample size for outcome analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03806231/Prot_SAP_000.pdf